CLINICAL TRIAL: NCT03284541
Title: A New Approach to Integrating Primary and Secondary HIV Prevention in Young Male Couples
Brief Title: Online HIV Prevention for Young Male Couples
Acronym: 2GETHER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Michael E. Newcomb, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DP2DA042417 (NIH)
Record Dates: First submitted 2017-06-23; First posted 2017-09-15 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Hiv; Chlamydia; Gonorrhea
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Chlamydia Infections; Gonorrhea

STUDY DESIGN:
Intervention Model Description: Couples are randomized into an experimental condition or control (existing public health practice).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2GETHER (Experimental): 2GETHER is an HIV prevention and relationship education program designed for young male couples. 2GETHER consists of 4 sessions (2 group sessions, 2 individualized couple session) administered over the course of 1 month (1 session per week). Group sessions focus on developing skills related to sexual health and relationship functioning, including HIV prevention in couples, communication skills, coping skills, problem-solving and acceptance. Individualized couple sessions focus on implementation of skills specific to the needs of each couple.
  Interventions: Behavioral: 2GETHER
- Existing Public Health Practice (Active Comparator): The control condition consists of the single-session Couples-Based HIV Counseling and Testing protocol for HIV-negative couples, the single-session Life-Steps medication adherence protocol for HIV-positive couples, or both intervention delivered jointly to serodiscordant couples
  Interventions: Behavioral: Existing Public Health Practice

INTERVENTIONS:
Behavioral: 2GETHER — Communication skills, coping skills, problem-solving, acceptance, HIV prevention
  Arms: 2GETHER
Behavioral: Existing Public Health Practice — HIV testing, medication adherence, HIV risk reduction
  Arms: Existing Public Health Practice

SUMMARY:
Young gay, bisexual, and other men who have sex with men (YMSM) are the only risk group in which rates of new HIV infections are on the rise. There has been a relative dearth of research dedicated to understanding these health disparities between gay/bisexual and heterosexual youth, and even less has focused on identifying factors that might promote resilience against negative health outcomes. Understanding both risk factors and processes of resilience is critical in developing efficacious interventions to improve health in this population.

Through a grant from the National Institutes of Health, the investigators completed formative research with young male couples. Qualitative interviews identified preferences for couples-based intervention format and content. While coupled YMSM expressed some interest in HIV prevention, they were most interested in building relationship skills. Coupled YMSM preferred group-based interventions in order to meet and learn from other couples but had concerns about discussing personal topics in groups. Quantitative analyses found that the rate of condomless sex in couples increased from adolescence to young adulthood. Further, the influence of older partners, partner violence, and drinking before sex were strongest in emerging adulthood. Informed by these, the investigators developed 2GETHER, which aims to reduce HIV transmission risk in couples by enhancing relationship functioning. 2GETHER is a four session program. The first two sessions are group sessions aimed at skills building, and the second two sessions are individualized couple sessions aimed at skills implementation. Modules address communication skills, coping with stress (both general and sexual minority-specific stress), relationship sexual satisfaction, and HIV transmission risk within the dyad and with outside partners. 2GETHER was designed to address HIV transmission risk in couples regardless of HIV status; couples learn to use behavioral and biomedical approaches to prevent both HIV acquisition (e.g., HIV testing, condom use, pre-exposure prophylaxis) and transmission (e.g., medication adherence to reduce viral load), with an overarching emphasis on the health of the couple.

The investigators completed a pilot trial of 2GETHER with funding from Northwestern University. The pilot trial enrolled 57 couples (N=114) and demonstrated feasibility, acceptability, and preliminary efficacy of 2GETHER. This pilot trial used a non-randomized pre-/post-test design because the goal was to evaluate feasibility, acceptability and preliminary effects in a large number of diverse couples to inform a future efficacy RCT. Post-test occurred 2 weeks post-intervention, or ~2 months post-baseline. The pilot trial recruited a diverse sample of couples in less than one year and each program module receive high ratings of acceptability during post-sessions evaluation and an exit interview. At the 2-week post-test, the investigators observed significant decreases in HIV risk behavior, improvements in motivation to reduce HIV risk, and improvements in relationship investment.

The current study will conduct a randomized controlled trial (RCT) to test the efficacy of 2GETHER, a novel couples-based intervention for young men who have sex with men (YMSM) that aims to reduce HIV transmission risk by optimizing relationship functioning. This RCT will be implemented online; both the experimental and control condition will be administered via video-conferencing technology to couples across the United States. The investigators will conduct this RCT with 200 dyads (total individual N=400), who will be randomized to receive the 2GETHER intervention or existing public health practice (PHP). PHP differs depending on the HIV status of individuals in the dyad. Couples in which both members are HIV-negative will receive the single-session Couples-Based HIV Counseling and Testing (CHCT) protocol. Couples in which both members are HIV-positive will receive the single session Life-Steps medication adherence protocol. Couples with discordant HIV statuses will receive both interventions jointly.

ELIGIBILITY:
Inclusion Criteria:

* Both members of the couple assigned male at birth and currently identify as male
* Both members of the couples at least 18 years of age; at least one between the ages of 18-29 years
* Both members of the couple identify one another as primary partners
* Couple has had oral or anal sex with one another in the past 3 months
* At least one member of the couple reports condomless anal sex with a serodiscordant or unknown status partner during the past 3 months
* At least one member of the couple reports an episode of binge-drinking or illicit drug use during the last 30 days
* Both members of the couple read and speak English at 8th grade level or better
* Both members have Internet access
* Both members audio recording of intervention sessions

Exclusion Criteria:

* Severe intimate partner violence during the past 3 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Both members of the dyad must be assigned male at birth and currently identify as male
Enrollment: 400 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Condomless anal sex | 12-months
  change in number of condomless anal sex acts with serodiscordant or unknown status partners
Occurrence of Sexually Transmitted Infections | 12-months
  the incidence (number of new cases or diagnoses) or Chlamydia and Gonorrhea at 12 months

SECONDARY OUTCOMES:
HIV Testing | Baseline, 3-, 6-, 9-, 12-months
  frequency of HIV testing among HIV-negative or unknown status participants
HIV Viral Load | Baseline, 12-months
  change in serum viral load among HIV-positive participants
Alcohol and Drug Use Problems | Baseline, 3-, 6-, 9-, 12-months
  change in problems associated with alcohol, marijuana and other illicit drug use
Relationship Satisfaction | Baseline, 3-, 6-, 9-, 12-months
  change in relationship satisfaction
Communication Skills | Baseline, 3-, 6-, 9-, 12-months
  change in communication skills with romantic partners

OTHER OUTCOMES:
Antiretroviral Medication Adherence | Baseline, 3-, 6-, 9-, 12-months
  change in ART medication adherence among HIV-positive participants
Pre-Exposure Prophylaxis | Baseline, 3-, 6-, 9-, 12-months
  initiation of pre-exposure prophylaxis among HIV-negative or unknown status participants
Pre-Exposure Prophylaxis Adherence | Baseline, 3-, 6-, 9-, 12-months
  change in pre-exposure prophylaxis adherence among participants have have initiated pre-exposure prophylaxis

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Newcomb, Ph.D., Principal Investigator — Northwestern University; Jim Carey, MPH, Study Director — Northwestern University; Ricky Hill, Ph.D., Study Director — Northwestern University
Locations (1):
- Northwestern University-Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sullivan PS, Salazar L, Buchbinder S, Sanchez TH. Estimating the proportion of HIV transmissions from main sex partners among men who have sex with men in five US cities. AIDS. 2009 Jun 1;23(9):1153-62. doi: 10.1097/QAD.0b013e32832baa34. PMID 19417579
- [Background] Greene GJ, Fisher KA, Kuper L, Andrews R, Mustanski B. "Is this normal? Is this not normal? There's no set example": Sexual Health Intervention Preferences of LGBT Youth in Romantic Relationships. Sex Res Social Policy. 2015 Mar;12(1):1-14. doi: 10.1007/s13178-014-0169-2. PMID 25678895
- [Background] Jiwatram-Negron T, El-Bassel N. Systematic review of couple-based HIV intervention and prevention studies: advantages, gaps, and future directions. AIDS Behav. 2014 Oct;18(10):1864-87. doi: 10.1007/s10461-014-0827-7. PMID 24980246
- [Background] Markman HJ, Rhoades GK. Relationship education research: current status and future directions. J Marital Fam Ther. 2012 Jan;38(1):169-200. doi: 10.1111/j.1752-0606.2011.00247.x. PMID 22283386
- [Background] Newcomb ME, Macapagal KR, Feinstein BA, Bettin E, Swann G, Whitton SW. Integrating HIV Prevention and Relationship Education for Young Same-Sex Male Couples: A Pilot Trial of the 2GETHER Intervention. AIDS Behav. 2017 Aug;21(8):2464-2478. doi: 10.1007/s10461-017-1674-0. PMID 28083833
- [Derived] Smith MS, Newcomb ME. Substance Use and Relationship Functioning Among Young Male Couples. Arch Sex Behav. 2023 Jul;52(5):2097-2110. doi: 10.1007/s10508-023-02627-1. Epub 2023 Jun 23. PMID 37351709
- [Derived] Newcomb ME, Swann G, Macapagal K, Sarno EL, Whitton SW, Mustanski B. Biomedical and behavioral outcomes of 2GETHER: A randomized controlled trial of a telehealth HIV prevention program for young male couples. J Consult Clin Psychol. 2023 Sep;91(9):505-520. doi: 10.1037/ccp0000823. Epub 2023 May 4. PMID 37141032
- [Derived] Newcomb ME, Sarno EL, Bettin E, Carey J, Ciolino JD, Hill R, Garcia CP, Macapagal K, Mustanski B, Swann G, Whitton SW. Relationship Education and HIV Prevention for Young Male Couples Administered Online via Videoconference: Protocol for a National Randomized Controlled Trial of 2GETHER. JMIR Res Protoc. 2020 Jan 27;9(1):e15883. doi: 10.2196/15883. PMID 32012111

DOCUMENTS (1):
  • Informed Consent Form (2019-03-04): https://cdn.clinicaltrials.gov/large-docs/41/NCT03284541/ICF_000.pdf